CLINICAL TRIAL: NCT00796640
Title: A Comparative Evaluation of the Pharmacokinetics and Pharmacodynamics Under Fasting and Fed Conditions of 2 Paliperidone Extended-release Pellet Formulations With Paliperidone Oral Solution in Healthy Adults
Brief Title: A Pharmacokinetics and Pharmacodynamics Study Under Fasting and Fed Conditions With Paliperidone Extended-release and Immediate-release Formulations
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CR004279
Record Dates: First submitted 2008-11-20; First posted 2008-11-24 (Estimated); Last update posted 2011-06-08 (Estimated); Status verified 2010-03

CONDITIONS: Schizophrenia
Keywords: Schizophrenia; Mood disorders; Antipsychotic drugs; ER Paliperidone
MeSH Terms: conditions — Schizophrenia; Mood Disorders

INTERVENTIONS:
Drug: ER Paliperidone

SUMMARY:
The purpose of this study is to compare the bioavailability of 2 extended release paliperidone pellet formulations under fasting and fed conditions with a 2 mg paliperidone oral solution under fasting conditions. Additional objectives are to compare the pharmacodynamic effects (postural changes in blood pressure and heart rate), to evaluate the safety and tolerability of each treatment, and to explore the relationship between CYP2D6 genotype and paliperidone exposure.

DETAILED DESCRIPTION:
This is a single-center, open-label, randomized, 5-way crossover Phase 1 study in non-smoking healthy men and women, aged between 18 and 55 years. The study consists of a screening period; a 5-way crossover, open-label treatment phase with 14 days washout between treatments; and end-of-study evaluations upon completion or at early withdrawal. Eligible volunteers will be randomly assigned to 1 of 5 treatment sequences. Each volunteer will receive the following treatments in random order: (A) paliperidone ER pellet formulation-1, as 1 capsule of 2.5 mg, under fasting conditions; (B) paliperidone ER pellet formulation-1, as capsule of 2.5 mg with food (high-fat breakfast); (C) paliperidone ER pellet formulation-2 as 1 capsule of 2.5 mg, under fasting conditions; (D) paliperidone ER pellet formulation-2 as 1 capsule of 2.5 mg with food (high-fat breakfast); (E) immediate release (IR) paliperidone oral solution, 2 mg (2 mL) of a 1-mg/mL solution, under fasting conditions. Alternative paliperidone ER formulations are being developed with the aim to increase bioavailability and reduce variability, without compromising the favorable effect on orthostatic hypotension as seen with ER OROS paliperidone. Therefore, in this study, the pharmacokinetics and pharmacodynamic properties, as well as the effect of food, of 2 alternative paliperidone ER pellet formulations will be investigated. Safety and tolerability will be monitored throughout the study.. Single doses of paliperidone ER pellet formulation-1, as 1 capsule of 2.5 mg, fasted; paliperidone ER pellet formulation-1, as 1 capsule of 2.5 mg with food (high-fat breakfast); paliperidone ER pellet formulation-2 as 1 capsule of 2.5 mg, fasted; paliperidone ER pellet formulation-2 as 1 capsule of 2.5 mg with food (high-fat breakfast); IR paliperidone oral solution, 2 mg (2 mL) of a 1-mg/mL solution, fasted.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (weight [kg]/height (m)²) range of 18.0 to 28.0 kg/m², inclusive
* Normotensive with supine (5 minutes) blood pressure between 100 and 140 mmHg systolic, inclusive, and diastolic between 60 and 90 mmHg, inclusive
* Healthy on the basis of a prestudy physical examination, medical history, electrocardiogram, and the laboratory results of blood biochemistry, hematology and urinalysis performed within 21 days before the first dose. If the results of the biochemistry, hematology or urinalysis testing are not within the laboratory's reference ranges the volunteer can be included only if the investigator judges that the deviations are not clinically significant. For liver function tests (alanine transaminase, aspartate transaminase, and bilirubin), the values must be contained within 2 times the upper limits of the normal laboratory reference ranges and for renal function tests, the values must be within the normal laboratory reference ranges
* Women must be postmenopausal for at least 1 year, surgically sterile, or practicing an effective method of birth control (e.g., prescription oral contraceptives, contraceptive injections, intrauterine device, double-barrier method, contraceptive patch, male partner sterilization and at the discretion of the investigator, total abstinence) before entry and throughout the study, as well as have a negative serum pregnancy test at screening. To ensure continued eligibility, women must have a negative urine test before each dose of study drug (Day -1 for each period).

Exclusion Criteria:

* Known allergy or history of significant hypersensitivity to heparin
* Recent history of alcohol or substance abuse. Test positive for the urine drug screen at screening or the urine drug screen or alcohol breath test at Day -1 for Period 1
* Relevant history of any cardiovascular, respiratory, neuropsychiatric, renal, hepatic, gastrointestinal (including surgeries, and malabsorption problems), endocrine, or immunologic diseases
* A decrease of greater than or equal to 20 mmHg systolic blood pressure 3 minutes after standing, or with symptoms of lightheadedness, dizziness or fainting upon standing at screening
* Positive result for any of the serology tests (hepatitis B, C and HIV)
* Have less than 1 bowel movement on average each day
* History of any cancer, with the exception of basal cell carcinoma
* History of smoking or use of nicotine-containing substances within the last 2 months, as determined by medical history and/or volunteer's verbal report. (Volunteers must agree to refrain from use throughout the study.)

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 35 (Actual)
Dates: Start 2003-09; Study Completion 2003-11 (Actual)

PRIMARY OUTCOMES:
To evaluate the pharmacokinetics of 2 ER pellet formulations of 2 mg-eq paliperidone in comparison to 2 mg IR paliperidone oral solution and to evaluate the effect of food on the pharmacokinetics of the ER pellet formulations

SECONDARY OUTCOMES:
To compare the pharmacodynamic effects of all treatments, to evaluate safety and tolerability as well as the relationship between genotypes (CYP2D6 and CYP3A4/5) and paliperidone exposure

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L. C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.

REFERENCES:
- See also: A pharmacokinetics and pharmacodynamics study under fasting and fed conditions with paliperidone extended-release and immediate-release formulations — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=578&filename=CR004279_CSR.pdf